CLINICAL TRIAL: NCT05359952
Title: Enhancing Clinical Communication About Sexual Health for Women With Gynecologic Cancer: Adaptation of a Multimedia Intervention
Brief Title: Women's Health Communication Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-1066
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Starting the Conversation (Experimental): Participants are asked to watch an educational video along with an accompanying workbook (called "Starting the Conversation"). Participants are also asked to review a list of resources about sexual and menopausal health relevant to gynecologic cancer.
  Interventions: Behavioral: Starting the Conversation; Behavioral: Sexual and Menopausal Health Resources Only
- Sexual and Menopausal Health Resources Only (Active Comparator): Participants are given the list of resources about sexual and menopausal health only.
  Interventions: Behavioral: Sexual and Menopausal Health Resources Only

INTERVENTIONS:
Behavioral: Starting the Conversation — The Starting the Conversation intervention consists of a brief educational video and accompanying workbook with activities to help prepare patients to discuss sexual and menopausal types of health concerns effectively with gynecologic cancer providers, including prioritizing concerns, tips for effective communication, communication practice, and self-feedback. In addition, participants receive a list of sexual and menopausal resources.
  Arms: Starting the Conversation
Behavioral: Sexual and Menopausal Health Resources Only — A list of resources on sexual/menopausal health both within and outside the institution, including websites.

SUMMARY:
The central goal of this randomized, controlled pilot study is to examine the feasibility, acceptability, and preliminary effects of an educational intervention (called "Starting the Conversation"; STC) on patient communication about sexual health in gynecologic cancer and other patient health outcomes. Approximately 30 women with a diagnosis of gynecologic cancer will be randomized to either participate in either the Starting the Conversation (STC) condition, consisting of an educational video, workbook, and list of resources on sexual and menopausal health, or to a control condition offering the resource guide only. Patients will be asked to review intervention materials prior to their next clinic visit with their gynecologic cancer provider. The investigators will examine effects of the interventions on patients' beliefs about communication about sexual health and on patients' communication about sexual health during clinic visits with their providers. Secondarily, the investigators will examine effects of the interventions on sexual outcomes and other health outcomes, including psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any stage (I-IV) gynecologic cancer (uterine, ovarian, cervical, vaginal/vulvar, fallopian tube, peritoneal)
* Receiving any treatment for gynecologic cancer or have completed acute treatment < 10 years ago
* Attending clinic visits in the course of follow-up care (i.e., not an initial consult visit)

Exclusion Criteria:

* Not able to speak English
* Eastern Cooperative Oncology Group (ECOG) Performance status score > 2
* Overt cognitive dysfunction or psychiatric disturbance or severe mental illness (e.g., dementia, suicidal behavior, or psychosis), as observed or judged by the researcher or referring source.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Started | 21 | 11
Completed | 20 | 11
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.5) | 65.4 (10.2) | 62.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 11 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 17 | 7 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 11 | 32
Education [Count of Participants; unit: Participants]
  High school or less | 3 | 2 | 5
  Some college | 4 | 4 | 8
  Completed college/graduate school | 14 | 5 | 19
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual/straight | 20 | 11 | 31
  Don't know | 1 | 0 | 1
Partnered Status [Count of Participants; unit: Participants]
  Married or partnered | 18 | 5 | 23
  Not partnered | 3 | 6 | 9
Disease Site [Count of Participants; unit: Participants]
  Endometrial | 11 | 6 | 17
  Ovarian | 8 | 3 | 11
  Cervical | 0 | 2 | 2
  Other | 2 | 0 | 2
Disease Stage [Count of Participants; unit: Participants] — Disease stage is based on tumor size, lymph node involvement, and presence of distant metastatic disease. Stages I-II are lower stage/better prognosis and stage IV is metastatic/worst prognosis.
  Participants
    Stage I-II | 10 | 8 | 18
    Stage III | 9 | 2 | 11
    Stage IV | 2 | 1 | 3
Primary Surgery [Count of Participants; unit: Participants]
  Hysterectomy/oophorectomy | 20 | 10 | 30
  None | 1 | 1 | 2
Chemotherapy Received [Count of Participants; unit: Participants]
  Chemotherapy received | 15 | 6 | 21
  No chemotherapy received | 6 | 5 | 11
Radiation Therapy Received [Count of Participants; unit: Participants]
  Radiation therapy received | 6 | 5 | 11
  No radiation therapy received | 15 | 6 | 21
Immunotherapy Received [Count of Participants; unit: Participants]
  Immunotherapy received | 9 | 4 | 13
  No immunotherapy received | 12 | 7 | 19
Hormonal Therapy Received [Count of Participants; unit: Participants]
  Hormonal therapy received | 1 | 3 | 4
  No hormonal therapy received | 20 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Enrollment
Description: Study enrollment, defined as the number of participants randomized out of the number of eligible patients approached for participation
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Study Candidates: All potentially eligible study candidates approached for participation.
Arm/Group | Study Candidates
Number analyzed (Participants) | 131
Participants | 32

2. Primary Outcome: Feasibility - Retention
Description: Number of enrolled participants that complete the final study survey.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 21 | 11
Participants | 20 | 11

3. Primary Outcome: Feasibility - Intervention Completion
Description: Number of participants randomized to receive the Starting the Conversation intervention who report having engaged at least somewhat with the video and/or accompanying workbook.
Time Frame: 2 weeks
Population: Only Starting the Conversation participants were asked about engagement with materials.
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 21 | 0
Participants
  Engaged with workbook and/or video | 21 |
  Did not engage with workbook or video | 0 |

4. Primary Outcome: Acceptability
Description: The number of participants randomized to receive the Starting the Conversation intervention who endorse at least 6 of 8 core components of the Starting the Conversation Intervention (defined as satisfaction with the intervention, informativeness of the intervention, helpfulness of the intervention, relevance of the intervention, ease of participation, approval of the intervention format, likelihood of recommending the intervention to others, and perceived importance of the intervention for people with gynecologic cancer).
Time Frame: 2 weeks
Population: Acceptability only measured in Starting the Conversation participants. One Starting the Conversation participant did not return the 2 week follow-up survey which measured acceptability.
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 0
Participants | 20 |

5. Secondary Outcome: Self-Efficacy - Post-Intervention
Description: Patients' confidence that they can discuss sexual concerns with their provider and ask their provider about sexual concerns. Scale ranges from 0-10, with higher scores indicating higher self-efficacy. Means will be reported.
Time Frame: 2 weeks
Population: One Starting the Conversation participant did not complete the 2-week follow-up assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
units on a scale | 8.18 [6.99 to 9.35] | 9.18 [8.15 to 10.22]

6. Secondary Outcome: Self-Efficacy - 2-Month Follow Up
Description: as for outcome 5
Time Frame: 2 months
Population: One Starting the Conversation participant did not complete the 2-month follow-up assessment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
units on a scale | 8.00 [6.59 to 9.41] | 8.68 [7.21 to 10.16]

7. Secondary Outcome: Clinical Communication - Discussion of Sexual Health
Description: Number of patients who discuss sexual health concerns in a clinic visit.
Time Frame: 2 weeks
Population: One Starting the Conversation participant did not complete the 2-week follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
Participants | 9 | 5

8. Secondary Outcome: Clinical Communication - Raising Topic of Sexual Health
Description: Number of patients who raise the topic of sexual health concerns in a clinic visit.
Time Frame: 2 weeks
Population: One Starting the Conversation participant did not complete the 2-week follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
Participants | 7 | 0

9. Secondary Outcome: Clinical Communication - Asking a Question About Sexual Health
Description: Number of patients who ask a question about sexual health concerns in a clinic visit.
Time Frame: 2 weeks
Population: One Starting the Conversation participant did not complete the 2-week follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
Participants | 9 | 3

10. Secondary Outcome: Change in Sexual Function
Description: Patients' self-reported sexual function will be measured using the 19-item Female Sexual Function Index (FSFI).Total scale scores range from 2 to 36, with higher scores indicating higher functioning. Positive mean change scores indicate increase in sexual functioning over time while negative mean change scores indicate decrease in sexual functioning over time.
Time Frame: baseline to 2 months
Population: One Starting the Conversation participant did not complete the 2-month follow-up assessment, and 6 Starting the Conversation participants did not have sufficient data on the scale to calculate a change score. Four Resources Only participants did not have sufficient data on the scale to calculate a change score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 14 | 7
score on a scale | 1.3 (3.9) | 4.5 (9.0)

11. Secondary Outcome: Sexual Activity
Description: A single item asking (yes/no) whether the participant had any kind of sexual activity in the past 30 days. Percent reporting sexual activity is reported.
Time Frame: 2 months
Population: One Starting the Conversation participant did not complete the 2-month follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
Participants | 10 | 4

12. Secondary Outcome: Psychological Distress - Depression
Description: Patients self-reported depression, as measured through depression subscale of the Hospital Anxiety & Depression Scale (HADS). The depression subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of depression. Means will be reported.
Time Frame: 2 months
Population: One Starting the Conversation participant did not complete the 2-month follow-up assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
score on a scale | 5.4 [3.45 to 7.35] | 4.55 [2.15 to 6.94]

13. Secondary Outcome: Psychological Distress - Anxiety
Description: Patients self-reported anxiety, as measured through anxiety subscale of the Hospital Anxiety & Depression Scale (HADS). The anxiety subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of anxiety. Means will be reported.
Time Frame: 2 months
Population: One Starting the Conversation participant did not complete the 2-month follow-up assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
Number analyzed (Participants) | 20 | 11
score on a scale | 8.20 [5.76 to 10.64] | 5.55 [2.87 to 8.22]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout study participation (2 months)
Arm/Group | Starting the Conversation | Sexual and Menopausal Health Resources Only
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 0/21 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT05359952/Prot_SAP_000.pdf